CLINICAL TRIAL: NCT03911882
Title: A Prospective, Open-label, Study to Evaluate the Efficacy and Tolerability of the Food Supplement CELERGEN in Patients With Fibromyalgia
Brief Title: Efficacy and Tolerability of CELERGEN in Fibromyalgia
Status: Completed | Type: Observational
Sponsor: Celergan SA (Industry)
Responsible Party: Sponsor
Other Study IDs: CELERGEN6007
Record Dates: First submitted 2019-03-25; First posted 2019-04-11 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-03

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Cytokines; TNF; Substance P; Spermine; Pain; Fatigue
MeSH Terms: conditions — Fibromyalgia; Pain; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Celergen Administration: The food supplement Celergen was administered to fibromyalgia patients following a protocol of a daily intake for the period of a total of 3 months (90 days)
  Interventions: Dietary Supplement: Celergen Administration

INTERVENTIONS:
Dietary Supplement: Celergen Administration — The food supplement Celergen was administered on a daily basis for a total of 3 months (90 days) to participating fibromyalgia patients

SUMMARY:
Celergén® is a dietary supplement with anti-inflammatory and antioxidant properties composed of marine sperm extract, hydrolyzed collagen, CoQ10, lutein and selenium. This is an open-label, prospective, study to evaluate the efficacy and tolerability of Celergen in 90 patients with Fibromyalgia. The study duration was 90 days and patients were evaluated by the: FIQ-R Fibromyalgia Impact Questionnaire Revised, Questionnaire of Health SF-12, Scale Clinical Global Impression Improvement assessed by the patient (PGI), and the Brief Pain Inventory (BPI). Blood samples were obtained at weeks 0 and 12 order for serum levels of Substance P and Tumor Necrosis Factor to measured blindly. Statistical analysis will be performed by analysis of variance for paired data.

DETAILED DESCRIPTION:
Fibromyalgia Syndrome (FMS) is a disease characterized by chronic widespread pain, along with muscle stiffness, sleep disorders, chronic fatigue, anxiety, depression, or neurocognitive deficiencies and autoimmune dysfunction. FMS prevalence is about 2% of the general population. Recently, a European study found a prevalence of 4.7% in all five countries surveyed, including Spain. The etiology of FMS is still unknown, but recent evidence supports the involvement of neuro-inflammation.

Celergén® is a dietary supplement with anti-inflammatory and antioxidant properties composed of a proprietory mixture of herring and mackerel milt semen and sperm-filled reproductive gland of male fish provided by Celergen Ltd, Luxemburg), hydrolyzed collagen, CoQ10, lutein and selenium.

This is an open-label, prospective, study to evaluate the efficacy and tolerability of Celergen in 90 patients with Fibromyalgia. The study duration was 90 days and patients were evaluated by the following:

INSTRUMENTS OF ASSESSMENT:

* Fibromyalgia Impact Questionnaire Revised (FIQR): The most commonly used scale to assess the severity and impact of fibromialgia.
* Brief Pain Inventory (BPI): Evaluates both pain intensity and interference with daily activities. The validated Spanish version will be used.
* Questionnaire of Health SF-12: This questionnaire, shortened version of the SF-36 version, has shown strong correlation with the latter both in relation to the physical and mental summary, presenting the advantage of its reduced complexity.
* Scale Clinical Global Impression Improvement assessed by the patient (PGI): A Likert scale of 7 points ranging from 1 (much better) to 7 (very much worse). It is used in most studies and clinical trials to assess the patients perception of the evolution of the disease in relation to the prescribed treatment.

COURSE OF STUDY:

The total duration of the study will be 12 weeks. Visit 1 (Week -0). - A general medical history, in which the possible diseases suffered by the patient and the medications they are taking for treatment is recorded, which should not be changed during the study. Data relating to previous or ongoing treatments (pharmacological or not) for FMS will also be collected. The inclusion and exclusion criteria will be checked, informed consent will be obtained. and blood will be drawn and stored at -80o C until the end of the study for biochemical analysis and comparison with blood drawn at the end of the study.

Visit 2 (baseline). - FIQR and the SF-12 and BPI questionnaires will be completed.

Celergen® treatment, to be administered as an adjunct to medication the patient is taking. A Celergen® capsule will be prescribed after breakfast, unmixed with taking other supplement or medication.

Visit 3 (Week 1). The FIQ, the BIS, the SF-12 and PGI questionnaires will be completed.

Visit 4 (Week 4). - Supplement tolerability will be assessed by recording the occurrence of adverse effects. The FIQ, the BIS, the SF-12 and PGI questionnaires will be completed.

Visit 5 (Week 8). - Supplement tolerability will be assessed by recording the occurrence of any adverse effects. The FIQ, the BIS, the SF-12 and PGI questionnaires will be completed.

Visit 6 (Week 12). - The FIQ, the BIS, the PGI, the SF-12 and PGI questionnaires will be completed. The end of the treatment will be recorded. Potential adverse reactions will be also be recorded. Final blood samples will be drawn for biochemical analysis.

STATISTICAL ANALYSIS:

Both the primary variable (the change in the initial and final mean scores of FIQ) and other quantitative variables (differences in mean scores on the BIS and SF-12) will be evaluated by analysis of variance for paired data.

Adverse reactions and PGI will be analyzed using descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with an established diagnosis of fibromyalgia according to the diagnostic criteria of the American College of Rheumatology of the year 2010.
* Patients who signed the informed consent to participate in the study

Exclusion Criteria:

* Patients suffering from any psychiatric disorder specified on Axis I DSM-IV- R other than major depression.
* Patients with a history or currently part of substance abuse.
* Patients who are pregnant or breastfeeding.
* Patients taking other dietary supplements with or without antioxidant character, or who are being treated with ozone therapy systemically.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Caucasian 18-60 years
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2016-04-29 (Actual); Primary Completion 2016-07-29 (Actual); Study Completion 2016-08-30 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire Revised | Compare values at T=week 1 (before treatment) with those at T=week 12 (end)
  Scale measuring overall fibromyalgia symptoms (0-100) For each symptom-based item (Questions 14 - 20) the raw score ranges from 0 to 10. If the patient marks between 2 hash marks the item is given a score that includes 0.5. Do Job: (Question 14) Raw score is final score. Pain: (Question 15) Raw score is final score. Fatigue: (Question 16) Raw score is final score. Rested: (Question 17) Raw score is final score. Stiffness: (Question 18) Raw score is final score. Anxiety: (Question 19) Raw score is final score. Depression: (Question 20) Raw score is final score. In each instance, the final score is the sum of the scores for the Physical Impairment, Feel Good, Pain, Fatigue, Rested, Stiffness, Anxiety, and Depression scales (does not include 2 work items.)
Brief Pain Inventory | Compare values at T=week 1 (before treatment) with those at T=week 12 (end)
  Scale measuring pain frequency and intensity (0-10) Brief Pain Inventory (Short Form) 2. On the diagram, shade in the areas where you feel pain. Put an X on the area that hurts the most.
  Yes No 0 1 2 3 4 5 6 7 8 9 10 0 1 2 3 4 5 6 7 8 9 10 0 1 2 3 4 5 6 7 8 9 10 4. Please rate your pain by marking the box beside the number that best describes your pain at its least in the last 24 hours. 6. Please rate your pain by marking the box beside the number that tells how much pain you have right now.
  0 1 2 3 4 5 6 7
Questionnaire of Health SF-12 | Compare values at T=week 1 (before treatment) with those at T=week 12 (end)
  Scale measuring quality of life (0-100) Choose one option for each questionnaire item.
  1. In general, would you say your health is:
  1. - Excellent
  2. - Very good
  3. - Good
  4. - Fair
  5. - Poor
  2. For how long (if at all) has your health limited you in each of the following activities?
  Limited for more than 3 months Limited for 3 months or less Not limited at all
  1. The kinds or amounts of vigorous activities you can do, like lifting heavy objects, running or participating in strenuous sports
     1 2 3
  2. The kinds or amounts of moderate activities you can do, like moving a table, carrying groceries, or bowling
     1 2 3
  3. Walking uphill or climbing a few flights of stairs
     1 2 3
  4. Bending, lifting, or stooping
     1 2 3
  5. Walking one block
     1 2 3
  6. Eating, dressing, bathing, or using the toilet
     1. 2 3 3. How much bodily pain have you had during the past 4 weeks:
     <!-- -->
     1. - None
     2. - Very mild
     3. - Mild
     4. - Moderate
Clinical Global Impression Improvement assessed by the patient (PGI) | Compare values at T=week 1 (before treatment) with those at T=week 12 (end)
  Scale measuring overall improvement (0-7) Severity scale The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Possible ratings are:[1]
  Normal, not at all ill Borderline mentally ill Mildly ill Moderately ill Markedly ill Severely ill Among the most extremely ill patients Improvement scale The Clinical Global Impression - Improvement scale (CGI-I) is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. and rated as:[1]
  Very much improved Much improved Minimally improved No change Minimally worse Much worse Very much worse

SECONDARY OUTCOMES:
Serum TNF level | Compare levels at T=1 week with levels at T=12 week
  ELISA measurement
Serum Substance P level | Compare levels at T=1 week 1 with levels at T=12 week
  ELISA measurement

CONTACTS AND LOCATIONS:
Overall Officials: Karin Freitag, Study Director — Clinica DFK, Madrid, Spain
Locations (1):
- Clinica DFK, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Catanzaro R, Celep G, Zerbinati N, Papacharalambous M, Nagpal R, Marotta F, Rastmanesh R, Milazzo M, Lorenzetti A, Bertuccelli G, Sollano J. In vitro protective effect of Celergen, a bioactive marine compound, on interleukin-6-related invasiveness of pancreatic cancer. Acta Biomed. 2014 May 9;85(1):44-51. PMID 24897969
- [Result] Catanzaro R, Zerbinati N, Solimene U, Celep G, Marotta F, Kushugulova A, Milazzo M, Tomella C, Bertuccelli G, Zhumadilov Z. Effect of Celergen, a marine derivative, on in vitro hepatocarcinogenesis. Drug Discov Ther. 2013 Oct;7(5):196-200. PMID 24270384
- [Derived] Tsilioni I, Pipis H, Freitag MSC, Izquierdo MDC, Freitag K, Theoharides TC. Effects of an Extract of Salmon Milt on Symptoms and Serum TNF and Substance P in Patients With Fibromyalgia Syndrome. Clin Ther. 2019 Aug;41(8):1564-1574.e2. doi: 10.1016/j.clinthera.2019.05.019. Epub 2019 Jul 11. PMID 31303280